CLINICAL TRIAL: NCT03300778
Title: A Randomised Controlled Trial of Aerobic Exercise for Adolescents With Subthreshold Depressive and/or Hypomanic Syndrome and for Non-clinical Adolescents
Brief Title: A Study of Aerobic Exercise for Adolescents With Subthreshold Mood Syndromes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Psychiatric Hospital (Other Government)
Responsible Party: Principal Investigator, Kangguang Lin, MD, PhD, Guangzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Guangzhou Brain Hospital
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Depressive Symptoms; Hypomania Nos Single Episode or Unspecified
Keywords: neurocognition; high-risk; prognosis
MeSH Terms: conditions — Depression | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercise (Experimental): Running at the intensity of 50%-70% of maximum heart rate (220-age) for 30 mins per day, 4 days per week, last for 3 months
  Interventions: Behavioral: aerobic exercise
- Placebo controlled group (Placebo Comparator): 6 sections of group activities: 3 sections of general psychological education; one section of group game, one section of group poetry reading activity, group singing entertainment.
  Interventions: Behavioral: Placebo controlled group

INTERVENTIONS:
Behavioral: aerobic exercise — Running at the intensity of 50%-70% of maximum heart rate (220-age) for 30 mins per day, 4 days per week, last for 3 months
  Arms: aerobic exercise
Behavioral: Placebo controlled group — 6 sections of group activities: 3 sections of general psychological education; one section of group game, one section of group poetry reading activity, group singing entertainment.
  Arms: Placebo controlled group

SUMMARY:
This study will investigate the effects of aerobic exercise on mental states, cognition, and long-term outcomes in adolescents with subthreshold depressive and/or hypomanic syndromes and in non-clinical school children

DETAILED DESCRIPTION:
Subthreshold depressive and hypomanic symptoms are common in adolescents, increasing the risk of developping into depression or bipolar disorder. Preliminary evidence shows that aerobic exercise might have positive effects in enhancing cognition and improving clinical symptoms in non-clinical and preclinical population and patients with mood disorders. This randomized controlled trial will investigate short-term (3 months) effects of aerobic exercise on cognition and clinical symptoms as well as the long-term (18 months) effects on the clinical outcomes of high-risk states.

ELIGIBILITY:
Inclusion Criteria:

1. 2 or more DSM-IV defined depressive symptoms, with one as core symptoms ( lost interest or pleasure in activity or depressed mood), lasting for 1 week.
2. 2 or more DSM-IV defined manic symptoms, last for 4 days, but falling short of the criteria for hypomania; or meeting DSM-5 defined symptoms criteria for hypomania, lasting 2-3 days.
3. non-clinical subjects

Exclusion Criteria:

* DSM-IV defined major depressive disorder
* DSM-IV defined hypo/mania
* History of or current other Axis I Disorders
* Diagnosed neurological or musculoskeletal disorder/injury,
* Uncontrolled cardiovascular or metabolic diseases that are not suitable for running
* Diagnosed hypertension
* Other diagnosed serious medical conditions that are not suitable for cycling
* Severe suicidal ideation
* Mental retardation
* Currently participating in a exercise program or activity, defined as 30 minutes of vigorous physical activity 4-5 times per week

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptoms | 12 weeks
  Changes in depressive symptoms measured by Patient Health Questionnaire (PHQ-9)
Changes in neurocognitive function | 12 weeks
  Changes in neurocognitive function measured by the MATRICS Consensus Cognitive Battery (MCCB) after three months (12 weeks) of aerobic exercise

SECONDARY OUTCOMES:
changes in anxious symptoms | 12 weeks
  anxious symptoms measured by Symptom Checklist 90 (SCL-90)
Changes in brain connectivity | 12 weeks
  using fMRI to measure brain connectivity
Number of participants with subthreshold mood symptoms | 18 months
  number of participants who meet the subthreshold syndromes for depression and/or hypomania
Changes in hypomanic symptoms | 12 weeks
  changes in hypomanic symptoms measured by Hypomania Check List-15(HCL-15)

CONTACTS AND LOCATIONS:
Overall Officials: kangguang Lin, MD; PhD, Principal Investigator — Guangzhou Brain hospital (Guangzhou Psychiatric Hospital); Guiyun Xu, MD, Study Director — Guangzhou Psychiatric Hospital
Locations (1):
- Guangzhou Brain Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided